CLINICAL TRIAL: NCT04489875
Title: Gum Chewing Reduces the Risk of Postoperative Ileus After Arthroplasty Procedures in The Elderly Population: A Parallel Design, Open-Label, Randomized Controlled Trial
Brief Title: Gum Chewing Reduces the Risk of Postoperative Ileus After Arthroplasty Procedures in The Elderly Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indus Hospital and Health Network (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ahsun Jiwani, Junior Biostatistician, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 456-784-9
Record Dates: First submitted 2020-06-01; First posted 2020-07-28 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Paralytic Ileus
Keywords: Hip Arthroplasty; Chewing gum; Sham Feeding
MeSH Terms: conditions — Intestinal Pseudo-Obstruction | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gum (Experimental): the patients in this arm will receive the post-operative oral feeding along with chewing gum which they'll be required to chew for at least 15 minutes before their meal 3 times a day
  Interventions: Behavioral: Chewing Gum
- No chewing gum (No Intervention): The patients in this arm will only receive the post-operative oral feeding

INTERVENTIONS:
Behavioral: Chewing Gum — The intervention would be chewing gum. The patients in the intervention arm would be asked to chew gum for 15 minutes before meals thrice a day.
  Arms: Chewing gum

SUMMARY:
Postoperative ileus (POI) is defined as a temporary cessation of bowel movement after a surgical procedure. Surgical procedures not only include abdominal or colorectal procedures but non-abdominal procedures as well. Cessation of bowel movement not only leads to disturbing constipation but also may lead to nausea, loss of appetite, and food intolerance. These patients tend to have more pain scores and dissatisfaction with the surgical management and team. The mechanism behind this condition is caused by a decrease in vagal parasympathetic stimulation. To break/prevent this mechanism, here comes the "sham feeding" (gum-chewing) effect where an increase in chewing and saliva enhances the gastric emptying and overall motility of gut as a cephalic phase of digestion even in non-gastro or colorectal surgeries. This effect is studied thoroughly in gastric, colorectal, and gynecological procedures. There is scarcity about its effect following orthopedic procedures specifically hip arthroplasty. The objective of this study is to assess the effect of adding gum-chewing to the conventional postoperative feeding regimen on restoring postoperative bowel function and length of stay in hospital of patients undergoing elective hip arthroplasty.

Interventions:

Behavioral intervention (Chewing gum) will be started the morning after surgery when the patient is fully awake and allowed to start taking an oral diet (which usually starts within 6-10 hours after surgery). In addition to the conventional postoperative feeding schedule, the patient will be given the gum to chew for at least 15 minutes each time, 3 times/day before the usual time of the meal, until the first flatus. The control group will have a conventional feeding schedule without chewing gum being added to their meals.

Hypothesis:

The investigators hypothesize that there is an association between gum chewing and the relief from postoperative ileus in hip arthroplasty patients.

Study Design:

Single-center, open-label, parallel design, superiority randomized-controlled trial with 2 treatment arms. The primary outcome will be the time interval in hours from the end of surgery until the passage of flatus, which is reported subjectively by the patient. The secondary outcome will be the time interval in hours from the end of surgery until the passage of stool. The other secondary outcome will be the postoperative hospital stay in days (surgery to discharge).

DETAILED DESCRIPTION:
Study Enrollment Procedures Enrollment will be a continuous process with screening and enrolling eligible patients admitted through the clinic electively for primary THR. Informed consent will be taken from the patient as per routine protocol before the arthroplasty procedures in the hospital. Research objectives, methodology, risks, and benefits will be explained in detail. Consent for the participation in the study will only be taken by the primary investigator at his clinic or the surgical resident on call preoperatively along with the consent for the surgical procedure.

Pre-Randomization Evaluations Screening The screening will involve the routine history taking and physical examination by the doctor and nursing staff in the clinic. Screening won't involve performing procedures that are not part of routine management. Special attention will be given on assessing the dental history and whether the patient is able to chew gum.

On-study/on-intervention evaluations After screening and eligibility, patients will be randomly allocated by a 1:1 ratio to the gum-chewing (gum) or control (no gum) groups using a computer-generated randomization sequence by the clinical trials unit (CTU), which they will provide to the PI, after patients' admission in the hospital. Patients will be followed from the time they reach the ward after surgery until their hospital discharge, which is usually around 7 days.

Data Collection:

Training of data collectors will be done by the PI to ensure the reliability and validity of the study. Data collectors will be recruited, preferably nurses or residents familiar with the hospital information management system (HIMS), the medical records and the CTU protocols. Training of data collectors will be done, and collectors will be strictly instructed to respect the autonomy of participants. Data collection will be done by the data collectors under the supervision of the PI and CTU. Questionnaires will be checked for consistency and logical data entries. Data entry will be done, and counter checked by the PI at regular intervals.

Data Storage:

Data collected will be coded and kept confidential without the identifiable information of patients. The confidentiality of the study participants will be maintained throughout the study period. Data collected will be kept confidential without identifiable information of patients who are identified by a number assigned. The hard copy forms will be retained in a secured location with the PI after data entry into computer software and will be kept as per hospital protocol. The password-protected drives will be used to store data with only the PI having access to it. The data will be available for AKU ethical review committee on request and might be published in a journal without disclosing any identifiable information of patients. Filled questionnaires will be stored for 5 years after the study is completed as per the policy of the institute.

Sample Size:

To the best of author's knowledge, this is the first research to study the effect of the gum-chewing post-arthroplasty procedure on time to flatus. Literature reported numerous studies on the same objective but only on post abdominal and colorectal surgery patients which gave minimum mean time to flatus post-surgery of 67 hours [3]. In arthroplasty, no handling of abdominal viscera is done, and the investigators assume the time of bowel return to function is considerably less. Hence, considering the rarity of previous literature and the number of cases to be operated in 6 months, investigators decided to recruit and study all the eligible patients during the study period from July 2020 to December 2020. The expected number of patients will be of 50 patients in each arm.

Plan of Analysis:

Statistical analysis will be done by using STATA software version 15. Mean ± SD will be computed for all the normally distributed quantitative variables. The median and interquartile range would be reported for the non-normally distributed quantitative variables. The categorical variables would be expressed in frequencies and percentages. Length of stay will be calculated by Kaplan-Meier analysis, with an unadjusted comparison of groups by mantel-cox log-rank test. Risk ratios for the time-to-become ileus free and time-to-discharge from the hospital will be calculated by cox proportional hazard regression model, considering the following independent variables: age, gender, operation type, diabetes mellitus, preoperative cardiovascular disease (ischemia /heart failure/dysrhythmias), PCA opiate use and presence/absence of chewing gum.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 50-70 years
* Undergoing elective primary hip arthroplasty surgery
* ASA grade I, II, and III
* The patients undergoing general anesthesia with/without neuraxial anesthesia

Exclusion Criteria:

* Patients refusing to consent
* Patients already having an established nasogastric (NG) tube/gastrostomy feeding, or unsafe/unable to swallow due to any neurological condition
* Patients with documented bowel disease other than peptic ulcers
* History of chronic constipation more than 3 days before surgery
* Inability to chew gum due to dental issues
* traumatic and revision cases of arthroplasty
* adjuvant surgical procedures (abdominal, thoracic, etc.) besides the primary arthroplasty procedure will also be excluded from the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Passage of Flatus | up to 12 hours post-operatively
  the time interval in hours from the end of surgery until the first passage of flatus, which is reported subjectively by the patient. Patients will be instructed to make note of the time when flatus is passed for the first time after surgery.

SECONDARY OUTCOMES:
passage of stool | up to 24 hours post-operatively
  the time interval in hours from the end of surgery until the first passage of stool, which is reported subjectively by the patient. Patients and the bedside nurse will be instructed to make note of the time when the stool is passed for the first time after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Obada Hassan, MSc. Epibio, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalyanwat as, jakhar m, jain s. Postoperative ileus: a study on the role of chewing gum to reduce its duration. Saudi surgical journal. 2018 jul 1;6(3):85.
- [Background] Begum s, shahzad n, murtaza g, rehman zu, hasnain zafar gc. Of post-operative ileus after colorectal surgeries: a randomized control trial. Clinics of sugery. 2018; 1 (1): 1-5. Age (years). 2018;55(13.5):51-9.
- [Background] Matros E, Rocha F, Zinner M, Wang J, Ashley S, Breen E, Soybel D, Shoji B, Burgess A, Bleday R, Kuntz R, Whang E. Does gum chewing ameliorate postoperative ileus? Results of a prospective, randomized, placebo-controlled trial. J Am Coll Surg. 2006 May;202(5):773-8. doi: 10.1016/j.jamcollsurg.2006.02.009. PMID 16648017
- [Background] van den Heijkant TC, Costes LM, van der Lee DG, Aerts B, Osinga-de Jong M, Rutten HR, Hulsewe KW, de Jonge WJ, Buurman WA, Luyer MD. Randomized clinical trial of the effect of gum chewing on postoperative ileus and inflammation in colorectal surgery. Br J Surg. 2015 Feb;102(3):202-11. doi: 10.1002/bjs.9691. Epub 2014 Dec 18. PMID 25524125
- [Background] Atkinson C, Penfold CM, Ness AR, Longman RJ, Thomas SJ, Hollingworth W, Kandiyali R, Leary SD, Lewis SJ. Randomized clinical trial of postoperative chewing gum versus standard care after colorectal resection. Br J Surg. 2016 Jul;103(8):962-70. doi: 10.1002/bjs.10194. Epub 2016 May 5. PMID 27146793
- [Result] Karmali S, Jenkins N, Sciusco A, John J, Haddad F, Ackland GL; POM-X Study Investigators. Randomized controlled trial of vagal modulation by sham feeding in elective non-gastrointestinal (orthopaedic) surgery. Br J Anaesth. 2015 Nov;115(5):727-35. doi: 10.1093/bja/aev283. Epub 2015 Aug 30. PMID 26323293
- [Result] Asao T, Kuwano H, Nakamura J, Morinaga N, Hirayama I, Ide M. Gum chewing enhances early recovery from postoperative ileus after laparoscopic colectomy. J Am Coll Surg. 2002 Jul;195(1):30-2. doi: 10.1016/s1072-7515(02)01179-1. PMID 12113542
- [Result] Noble EJ, Harris R, Hosie KB, Thomas S, Lewis SJ. Gum chewing reduces postoperative ileus? A systematic review and meta-analysis. Int J Surg. 2009 Apr;7(2):100-5. doi: 10.1016/j.ijsu.2009.01.006. Epub 2009 Jan 31. PMID 19261555
- [Derived] Hasan O, Mazhar L, Jiwani A, Begum D, Lakdawala R, Noordin S. Gum Chewing, Added to Conventional Feeding, Reduces Risk of Post-Operative Ileus after Elective Hip and Knee Arthroplasty Procedures in Elderly Population: A Protocol for a Parallel Design, Open-Label, Randomized Controlled Trial. Int J Surg Protoc. 2021 Aug 9;25(1):165-170. doi: 10.29337/ijsp.158. eCollection 2021. PMID 34435165